CLINICAL TRIAL: NCT03954314
Title: Decreasing Postoperative Blood Loss by Topical vs. Intravenous Tranexamic Acid in Open Cardiac Surgery (DEPOSITION) Study
Brief Title: DEPOSITION - Decreasing Postoperative Blood Loss by Topical vs. Intravenous Tranexamic Acid in Open Cardiac Surgery
Acronym: DEPOSITION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Upon the Data Safety Monitoring Board review of the interim analysis (75% of participants have finished their follow-up) on November 17, 2023, they made a recommendation to stop recruitment into the trial.
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEPOSITION
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Bleeding; Surgical Blood Loss; Seizures
Keywords: Tranexamic Acid; On-pump Cardiac Surgery
MeSH Terms: conditions — Hemorrhage; Blood Loss, Surgical; Seizures | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Tranexamic Acid intravenous + Placebo topical versus Placebo intravenous + Tranexamic Acid topical
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacy will prepare 2 syringes of 50 ml of topical TxA (5 g) or placebo. They will also prepare for the same patient 2 syringes of 50 ml (5 g) for intravenous (i.v.) injection or placebo. TxA is similar in all aspects to normal saline. Blinding of both teams will be easy. The syringes will be prepared and randomized in pharmacy before the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Tranexamic Acid/Placebo (Active Comparator): Topical Tranexamic Acid 5g to 10g (50 to 100mL) or placebo. The topical will be poured into the pericardial and mediastinal cavities after protamine administration.
  Interventions: Drug: Tranexamic Acid
- Intravenous Tranexamic Acid/Placebo (Active Comparator): Intravenous Tranexamic Acid 1 to 10g (10 to 100mL) or placebo administered intravenously at the induction of anesthesia as a bolus-infusion.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic Acid is a medication used to treat or prevent excessive blood loss from major trauma, post partum, surgery, tooth removal, nose bleeds, and heavy menstruation.
  Other Names: Cyklokapron

SUMMARY:
The aim is to conduct a double-dummy multi-centre randomized controlled clinical trial of application of topical dose of tranexamic acid (TxA) versus the usual intravenous TxA in patients undergoing on-pump cardiac surgery.

DETAILED DESCRIPTION:
Postoperative bleeding related to open cardiac surgery increases the rates of complications and mortality. It results from the blood thinners that are needed for use. Intravenous tranexamic acid (TxA) has become a mainstay in cardiac surgical procedures for decreasing bleeding and minimizing transfusion requirements. Although intravenous TxA is usually well tolerated, there is a well-known risk (1 to 4%) of postoperative seizures. This is due to the similarity between TxA and the brain tissues. The aim is to eliminate the risk of seizures but to maintain the protection against bleeding. When TxA is used directly on the tissues (topically) for other type of surgeries (joints), TxA is effective to reduce blood loss and transfusions. The aim is to prove that direct application of TxA on the heart can eliminate postoperative seizures and reduce the amount of blood transfusions in patients who have cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Undergoing a cardiac surgical procedure (i.e. isolated coronary artery bypass graft (CABG), isolated single cardiac valve surgery or a combination of both or isolated ascending aorta replacement) with the use of cardiopulmonary bypass (CPB) and median sternotomy
3. Provide written informed consent

Exclusion Criteria:

1. Allergy to tranexamic acid
2. Undergoing minimally invasive surgery
3. Fulfill any of the following transfusion risk factors (A-D):

   A. Emergency surgery B. History of bleeding disorder C. Inherited thromboembolic or hemorrhagic disease D. Infective endocarditis (active)
4. History of previous cardiac surgery
5. Estimated glomerular filtration rate <30 mL/min (CKD-EPI equation) or on dialysis
6. Pre-operative hemoglobin > 170 g/L or <110 g/L
7. Pre-operative thrombocytopenia (<50,000 platelets per µL)
8. Expected circulatory arrest
9. Pregnancy or breast feeding
10. Previously enrolled in the DEPOSITION trial
11. Refusal of blood products
12. Pericardiectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3242 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
The proportion of patients experiencing an in-hospital seizure | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  To determine in patients undergoing on-pump cardiac surgery, if topical tranexamic acid (intra-pericardial) is superior to the usual intravenous tranexamic acid administration for reducing the risk of in-hospital seizure.

SECONDARY OUTCOMES:
The proportion of patients in-hospital who receive red blood cell transfusions | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  To determine in patients undergoing on-pump cardiac surgery, if topical tranexamic acid (intra-pericardial) compared with intravenous tranexamic acid administration is associated with a non-inferior risk of in-hospital red blood cell transfusion.

OTHER OUTCOMES:
Blood product transfusions | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  Analyzed using an ANCOVA model. In such a model, bags of blood product will be included as a dependent variable, whereas dose of tranexamic acid and treatment will be included as covariates.
Re-operation for bleeding or tamponade | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  Analyzed with a binomial regression
Duration of ICU stay | Number of hours in ICU are being collected at the Post-Operative Visit. Hour collection will start upon arrival at ICU post surgery and stop at ICU exit, up to 10 days maximum.
  Analyzed using an ANCOVA model.
MACE (Death, non-fatal Myocardial Infarction (MI), or non-fatal stroke) | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  A Cox proportional hazard model will be used to analyze the time to the first occurrence of the composite of death, non-fatal MI, or non-fatal stroke (MACE).

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lamy, MD, Principal Investigator — Population Health Research Institute
Locations (16):
- Canada (8):
  - Kelowna General Hospital, Kelowna, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Hamilton Health Sciences - General Hospital, Hamilton, Ontario
  - CHUM, Montreal, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CIUSSS NIM/Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - IUCPQ, Québec, Quebec
- China (2):
  - Beijing Anzhen Hospital, Beijing
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
- Nemocnice Agel Třinec, Třinec, Czechia
- University of Malaya, Kuala Lumpur, Malaysia
- Auckland City Hospital, Auckland, New Zealand
- Russia (3):
  - Petrovsky National Research Centre, Moscow
  - E.Meshalkin National Medical Research Center, Novosibirsk
  - Saint-Petersburg State University Hospital, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spence J, Long S, Tidy A, Raymer K, Devereaux PJ, Lamy A, Whitlock R, Syed S. Tranexamic Acid Administration During On-Pump Cardiac Surgery: A Survey of Current Practices Among Canadian Anesthetists Working in Academic Centers. Anesth Analg. 2017 Dec;125(6):1863-1870. doi: 10.1213/ANE.0000000000002422. PMID 28858904
- [Background] Lamy A, Tong W, Gao P, Chrolavicius S, Gafni A, Yusuf S, Connolly SJ. The cost of clopidogrel use in atrial fibrillation in the ACTIVE-A trial. Can J Cardiol. 2012 Jan-Feb;28(1):95-101. doi: 10.1016/j.cjca.2011.08.112. Epub 2011 Oct 8. PMID 21983111
- [Result] Habbab LM, Hussain S, Power P, Bashir S, Gao P, Semelhago L, VanHelder T, Parry D, Chu V, Lamy A. Decreasing Postoperative Blood Loss by Topical vs. Intravenous Tranexamic Acid in Open Cardiac Surgery (DEPOSITION) study: Results of a pilot study. J Card Surg. 2019 May;34(5):305-311. doi: 10.1111/jocs.14027. Epub 2019 Mar 25. PMID 30908754
- [Result] Myles PS, Smith JA, Forbes A, Silbert B, Jayarajah M, Painter T, Cooper DJ, Marasco S, McNeil J, Bussieres JS, McGuinness S, Byrne K, Chan MT, Landoni G, Wallace S; ATACAS Investigators of the ANZCA Clinical Trials Network. Tranexamic Acid in Patients Undergoing Coronary-Artery Surgery. N Engl J Med. 2017 Jan 12;376(2):136-148. doi: 10.1056/NEJMoa1606424. Epub 2016 Oct 23. PMID 27774838
- [Result] Fergusson DA, Hebert PC, Mazer CD, Fremes S, MacAdams C, Murkin JM, Teoh K, Duke PC, Arellano R, Blajchman MA, Bussieres JS, Cote D, Karski J, Martineau R, Robblee JA, Rodger M, Wells G, Clinch J, Pretorius R; BART Investigators. A comparison of aprotinin and lysine analogues in high-risk cardiac surgery. N Engl J Med. 2008 May 29;358(22):2319-31. doi: 10.1056/NEJMoa0802395. Epub 2008 May 14. PMID 18480196
- [Result] Mazer CD, Whitlock RP, Fergusson DA, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, Carrier FM, McGuinness S, Young PJ, Byrne K, Villar JC, Royse A, Grocott HP, Seeberger MD, Mehta C, Lellouche F, Hare GMT, Painter TW, Fremes S, Syed S, Bagshaw SM, Hwang NC, Royse C, Hall J, Dai D, Mistry N, Thorpe K, Verma S, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Six-Month Outcomes after Restrictive or Liberal Transfusion for Cardiac Surgery. N Engl J Med. 2018 Sep 27;379(13):1224-1233. doi: 10.1056/NEJMoa1808561. Epub 2018 Aug 26. PMID 30146969
- [Result] Kalavrouziotis D, Voisine P, Mohammadi S, Dionne S, Dagenais F. High-dose tranexamic acid is an independent predictor of early seizure after cardiopulmonary bypass. Ann Thorac Surg. 2012 Jan;93(1):148-54. doi: 10.1016/j.athoracsur.2011.07.085. Epub 2011 Nov 4. PMID 22054656
- [Derived] Lamy A, Sirota DA, Jacques F, Poostizadeh A, Noiseux N, Efremov S, Demers P, Akselrod B, Wang CY, Arora RC, Branny P, McGuinness SP, Brown CD, Jeanmart H, Zhao Q, Zhang H, Belley-Cote EP, Whitlock RP, Browne A, Copland I, Vincent J, Khatun R, Balasubramanian K, Bangdiwala SI, McGillion MH, Fox-Robichaud AE, Spence J, Yusuf S, Devereaux PJ; DEPOSITION Study Group. Topical Versus Intravenous Tranexamic Acid in Patients Undergoing Cardiac Surgery: The DEPOSITION Randomized Controlled Trial. Circulation. 2024 Oct 22;150(17):1315-1323. doi: 10.1161/CIRCULATIONAHA.124.069606. Epub 2024 Apr 8. PMID 38587333